CLINICAL TRIAL: NCT05610670
Title: Access to Parenthood and Gynecological Follow-up After Organ Transplantation
Acronym: FerGyTransplan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_0181
Record Dates: First submitted 2022-10-10; First posted 2022-11-09 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Parenthood Status; Transplant Lung; Transplant Kidney
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients who underwent a kidney/pulmonary transplant before the age of 40 (Other): The questionnaire will allow us to complete the information not obtained from the patients' files on the one hand, and to collect their experiences regarding the desire and/or achievement of a pregnancy, but also their gynecological follow-up in the broad sense, on the other hand.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire will allow us to complete the information and to collect their experiences regarding the desire and/or achievement of a pregnancy, but also their gynecological follow-up in the broad sense, on the other hand.

SUMMARY:
Solid organ transplants affect subjects of all ages, including young women of childbearing age. The improvement in the management of young female transplant patients makes it possible to consider pregnancies, about which the literature reports reassuring data on small series. The question of gynecological follow-up, access to parenthood, as well as the information and experience of patients regarding these issues after transplantation have thus become topical issues.

DETAILED DESCRIPTION:
Nowadays, solid organ transplantation is a common procedure performed all over the world on patients of all ages. It represents about 900,000 procedures per year worldwide and a little over 6,100 in France (who.int). It has become indispensable for treating certain pathologies: for example, renal transplantation is the best alternative for treating end-stage renal failure, both from the point of view of effectiveness and medical benefit for the patient and from an economic standpoint. As the indications are increasingly broad, the Foch Hospital is the leading French center for lung transplantation mainly on patients with cystic fibrosis but recently transplanted a lung on a patient with end-stage respiratory failure due to Covid-19.

Patients who have undergone a solid organ transplantation require, after the procedure and more generally throughout their life, a global management by a multidisciplinary team in order to maintain a regular and adapted surveillance, in particular because of the immunosuppressive treatments, which are subject to numerous complications (benefit-risk balance between the rejection episodes and the infectious and carcinological risks).

Pregnancy adds an increased risk of morbidity for transplant patients of childbearing age. However, progress in terms of follow-up and post-transplant treatment increasingly allows them to be authorized. In the literature, there are already some reassuring series on the course of pregnancies after renal or pulmonary transplantation, but the studies are very often limited to strict obstetrical and neonatal criteria.

Moreover, the risk of cervical dysplasia is increased in transplant patients. While the HAS recommends "joint and close follow-up between the referring physician and the gynecologist", the gynecological follow-up of young women after solid organ transplantation does not meet any specific recommendation at present.

Finally, the question of parenthood has a major place in our societies. It is in this context that it seems interesting to us to look at the gynecological follow-up of transplant patients by integrating pregnancies and their outcomes, but also the patients' experiences with regard to their desire for parenthood.

ELIGIBILITY:
Inclusion Criteria:

* Women treated at the Foch Hospital for kidney/pulmonary transplantation or for kidney transplantation at the Bicêtre Hospital from 2010 to 2018 (lung) and 2019 (kidney)
* Having been transplanted before the age of 40
* Over 18 years of age
* Have signed a consent form
* Affiliated to a health insurance plan

Exclusion Criteria:

* Transplantectomy within 1 year (kidney) or 2 years (lung) of transplantation
* Be deprived of liberty or under guardianship
* Not speaking or understanding French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 116 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 1 month after inclusion
  Pregnancy rate (defined as the number of confirmed pregnancies (positive urine or plasma pregnancy test) out of the number of patients with a pregnancy desire) and obstetrical outcomes in renal/pulmonary transplant patients with a pregnancy desire

SECONDARY OUTCOMES:
Gynecological evaluation post-transplant | 1 month after inclusion
  Frequency of gynecological follow-up, date of return of cycles, evaluation of contraception and occurrence of post-transplant cervical dysplasia
Satisfaction with information received regarding the risks of post-transplant pregnancy | 1 month after inclusion
  Satisfaction with information received regarding the risks of post-transplant pregnancy prior to transplantation on a scale of 1 to 5 (1 : not good at all - 5 : very good)
Patients' experience | 1 month after inclusion
  patients' experience of their parental project and the support of the medical team in the event of difficulties in accessing parenthood (scale from 1 to 5, 1 : not good at all - 5 : very good).
Conception time | 1 month after inclusion
  Conception time
use of MPA | 1 month after inclusion
  number of participants who used of MPA

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No